CLINICAL TRIAL: NCT05432557
Title: External Oblique Intercostal Plane Block Versus Subcostal Transversus Abdominis Plane Block in Supra-umbilical Surgical Incisions; Randomized Controlled Double Blinded Clinical Trial
Brief Title: External Oblique Intercostal Plane Block Versus Subcostal Transversus Abdominis Plane Block in Supra-umbilical Surgical Incisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Samar Rafik Mohamed Amin, lecturer of anesthesia and surgical ICU, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC 1-5-2022
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group E (Experimental): patients will receive ultrasound guided external oblique intercostal plain block.
  Interventions: Procedure: external oblique intercostal plain block (EOIP)
- Group T (Experimental): patients will receive ultrasound guided subcostal transversus abdominis plane block.
  Interventions: Procedure: subcostal transversus abdominis plane block (SCTAP)
- Group C (Placebo Comparator): patients won't receive LA injection
  Interventions: Other: control group

INTERVENTIONS:
Procedure: external oblique intercostal plain block (EOIP) — A high-frequency linear ultrasound probe will be placed in a longitudinal parasagittal orientation at the sixth intercostal space in the anterior midaxillary line. A 21G 10 cm needle will be inserted using an in plane approach. The tip of the needle will be placed into the fascial plane on the deep aspect of the external oblique muscle. A volume of 20 mL of LA mixture (10 mL of bupivacaine 0.5%, 5 mL of lidocaine 2% and 5 mL of normal saline to make a mixture totaling 20 ml.) will be injected.
  Arms: Group E
Procedure: subcostal transversus abdominis plane block (SCTAP) — The US probe will be placed immediately below the costal margin on oblique plane toward the lateral close to midline to identify the rectus abdominis muscle. The transversus abdominis muscle will be identified lying posterior to the rectus muscle. An 8cm 22-gauge block needle will be inserted using an in- plane approach. transversus abdominis plane will be accessed by placing the needle adjacent to costal margin but medial to linea semilunaris. The needle will be advanced slowly in-plane to promote hydrodissection along the oblique subcostal line. A volume of 20 mL of LA mixture (10 mL of bupivacaine 0.5%, 5 mL of lidocaine 2% and 5 mL of normal saline to make a mixture totaling 20 ml.) will be injected.
  Arms: Group T
Other: control group — No LA injection
  Arms: Group C

SUMMARY:
Various newer techniques have been proposed to enhance analgesia in upper abdominal region. The subcostal transverse abdominis plane (SCTAP) block is the deposition of local anesthetic in the transverse abdominis plane inferior and parallel to the costal margin. There is a growing consensus that the SCTAP block provides better analgesia for upper abdominal incisions than the traditional transverse abdominis plane block.

The External oblique intercostal plane (EOIP) block is a novel technique reported by Hamilton et al. performed EOPB by administering LA superior or deep of the external oblique muscle from the sixth intercostal space leading to the blockage of thoracoabdominal nerves at T6-T10. It has several attractive aspects such as easy sono-anatomy ribs one strip of muscle so easy to demonstrate even in obese patients, there is a bony backstop, easy expandable fascial plane that can accommodate a catheter and it is shallow block with no big vessels nearby.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status grade I -II,
2. Scheduled to undergo elective supra-umbilical surgeries under GA (epigastric herniotomy- gastrectomy- open cholecystectomy- nephrectomy).

Exclusion Criteria:

1. Allergy to local anesthetics,
2. Infection at the site of injection,
3. Coagulopathy,
4. Chronic pain syndromes,
5. Prolonged opioid medication,
6. Patients who received any analgesic 24 h before surgery.
7. Chronic liver disease, chronic renal disease, and cognitive impairment.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
amount of postoperative morphine consumed | 24 hours postoperatively
First postoperative analgesics request | 24 hours postoperatively

SECONDARY OUTCOMES:
Postoperative pain score | at 1, 2,4 , 8, 16 and 24 hours postoperatively
  pain evaluated by VAS (visual analogue score).
Incidence of Postoperative nausea & vomiting (PONV) | 24 hours postoperatively
  Number of patients developing PONV
incidence of complications related to the block | 24 hours postoperatively
  agitation, dizziness, tinnitus, tremors, and numbness.

CONTACTS AND LOCATIONS:
Locations (1):
- Samar Rafik Amin, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No